CLINICAL TRIAL: NCT03189680
Title: A High-Intensity Multi-Component Agility Intervention Improves Parkinson's Patients' Clinical and Motor Symptoms
Brief Title: Agility Training in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Somogy Megyei Kaposi Mór Teaching Hospital (Other)
Collaborators: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Tollár József, Principal investigator, Somogy Megyei Kaposi Mór Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IKEB0012/2015
Record Dates: First submitted 2017-05-31; First posted 2017-06-16 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2017-06

CONDITIONS: Parkinson Disease
Keywords: sensorimotor training; exergaming; posture; quality of life
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: The single-arm, 3-week-long intervention, administered daily, targeted postural instability and mobility using at-limit intensity sensorimotor and visuomotor agility training (n = 35, 17 males) conceptualized but seldom implemented previously. Each of the 15 training sessions lasted 60 minutes. Patients performed each exercise under increasingly difficult conditions and speed according to principles of periodization. All patients kept an exercise log detailing the positive and negative effects of the intervention on clinical and motor symptoms. The logs and attendance were checked daily. The no-intervention control, consisting of PD patients (n = 20, 12 males) received unsupervised standard care, consisting of the prescribed medications and daily, unsupervised 30 minutes of exercises at home.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise therapy (Experimental): Parkinson's disease group that receive 3 weeks of intensive exercise therapy in a rehabilitation center.
  Interventions: Other: Exercise therapy
- Control (No Intervention): Parkinson's disease control group that will not receive exercise treatment.
- Healthy (No Intervention): A healthy group whose results will be compared with Parkinson's disease groups.

INTERVENTIONS:
Other: Exercise therapy — 3-week-long intervention, administered daily, targeted postural instability and mobility using at-limit intensity sensorimotor and visuomotor agility training
  Other Names: Control
  Arms: Exercise therapy

SUMMARY:
To determine the effects of an unusually highly intensity and individualized sensorimotor and visuomotor agility exercise program on non-demented PD patients' clinical symptoms, mobility, and postural stability.

DETAILED DESCRIPTION:
Design: Intervention study

Setting: Outpatient rehabilitation center

Participants: 55 Parkinson's disease (PD) patients completed the trial and 42 serves as comparison healthy controls

Intervention: An initial screening established specific dysfunctions of PD patients with Hoehn-Yahr stage 2-3 who were then randomly assigned to standard care (n = 20) or standard care plus at-limit intensity, individualized agility program (15 sessions, 3 weeks, n = 35).

Main outcome measures: Movement Disorder Society Unified Parkinson Disease Rating Scale, Motor Experiences of Daily Living, a measure sensitive to changes in a broad spectrum of PD symptoms

In group time, repeated measurements of variance analysis were compared to the picture parkinson's disease based on MDS-UPDRS M-EDL, Beck depression score, PDQ-39, EQ5D VAS, Schwab & England scale. The TUG test and 12 static posturographic measurements are compared and compared to the healthy group as a standard.

An at-limit and individualized sensorimotor and visuomotor agility exercise program vs. standard care, will improve non-demented, stage 2-3 PD patients' clinical symptoms, mobility, and postural stability by functionally meaningful margins.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease
* Hoenh Yahr scale of 2-3
* Instability problem

Exclusion Criteria:

* Severe heart problems
* Severe demeanor
* Alcoholism
* Drug problems

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-05-11 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
EQ5D-5L | 0-5 scale (3 week-long, higher number is better)
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Somogy Megyei Kaposi Mór Teaching Hospital, Kaposvár, Somogy County, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886
- [Derived] Tollar J, Nagy F, Kovacs N, Hortobagyi T. Two-Year Agility Maintenance Training Slows the Progression of Parkinsonian Symptoms. Med Sci Sports Exerc. 2019 Feb;51(2):237-245. doi: 10.1249/MSS.0000000000001793. PMID 30303934
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/